CLINICAL TRIAL: NCT01787617
Title: Aerobic Plus Resistance Training and Insulin Sensitivity in African American Men
Acronym: ARTIIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 11038
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: Exercise Training; Strength Training; African American Men; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): We will randomly assign 52 individuals to a no exercise healthy living group.
  Interventions: Behavioral: Control Group
- Aerobic Plus Resistance Training Group (Experimental): We will randomly assign 52 individuals to an aerobic plus resistance training group.
  Interventions: Behavioral: Aerobic Plus Resistance Training Group

INTERVENTIONS:
Behavioral: Aerobic Plus Resistance Training Group — Participants randomized to this intervention will engage in both aerobic and resistance training in accordance with Physical Activity Guidelines for Americans, that is 150 minutes of aerobic training and 2 days of additional 20 minutes of resistance training. The aerobic training component will be completed on a treadmill and target training intensity will be self-selected at 65% to 85% of maximal aerobic capacity. Each resistance training session will consist of both upper and lower body exercises: 2 sets of 9 exercises with each set consisting of 10 repetitions.
  Other Names: Exercise
  Arms: Aerobic Plus Resistance Training Group
Behavioral: Control Group — Participants randomized into the control group will not be provided with memberships to any exercise facility, nor will they receive behavioral instruction on how to increase physical activity. They will receive information on living a healthy lifestyle. Such minimal interventions have not been shown to increase physical activity in participants. The participants in this group will undergo the baseline, 10 week, and 20 week testing.
  Other Names: Healthy Living
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the effect of an exercise training intervention on the ability of African American males to use insulin properly. Insulin is a hormone that helps the body use glucose.

DETAILED DESCRIPTION:
This study is designed to assess the effect of exercise training on insulin resistance in African American males. African American males have higher rates of diabetes and lower levels of fitness when compared to Caucasian males. A project such as this is necessary because there is evidence to show that exercise training can reduce the risk of developing diabetes, though no studies have been conducted in African American males. In addition, ARTIIS will test the effect adhering to the 2008 Physical Activity Guidelines for Americans (150 minutes of moderate intensity aerobic activity and 2 days of 20 minutes of muscular strength activity), on insulin resistance in African American men. This study will provide important information that can either strengthen or refine current physical activity recommendations. Furthermore, this intervention will be delivered through community facilities in order to increase the likelihood that the intervention will be sustainable.

ELIGIBILITY:
Inclusion Criteria:

* You completed the three run-in screening visits.
* You self-identify as a male of African descent.
* You are 35 to 70 years of age.
* You have a BMI (ratio of your height to your weight) greater than or equal to 25.0 kg/m2 and less than or equal to 40 kg/m2.
* You have a family history of diabetes.
* You are not currently physically active for 20 minutes each time for 3 or more days per week for the last 6 months. You are not participating in regular muscle building exercise.
* You are willing to give informed consent, willing to be randomized to either the healthy living intervention group or the aerobic plus resistance training exercise group, and willing to follow the protocol for the group to which you have been assigned.

Exclusion Criteria:

* You drink more than 14 alcoholic drinks per week.
* You plan to move out of the study area within the next 6 months, or plan to be out of the study area for more than 4 weeks during the course of the study.
* You have another member of your household participating in the study.
* You have serious health conditions that would interfere with the intervention goals
* History of cardiovascular disease (CVD) or disorders and are not under the care of a physician to treat the condition, or fail to provide written documentation from your physician indicating that the physician approves of your entering the study
* Have high blood pressure (greater than 155/99 mmHg) and are not under the care of a physician to treat the condition or fail to provide written documentation from your physician indicating that the physician approves of your entering the study
* Have a previous diagnosis of diabetes (Type 1 or 2) or a fasting plasma glucose of >125 mg/dl
* Have elevated bad cholesterol (greater than or equal to 190mg/dl) or triglycerides (great than or equal to 300) and are not under the care of a physician to treat the condition or fail to provide written documentation from your physician indicating that the physician approves of you entering the study
* Are currently taking medications for diabetes or chronic steroid use
* Have chronic or recurrent respiratory, gastrointestinal, neuromuscular, neurological or psychiatric conditions
* Have had cancer requiring treatment in the past 5 years, expect for non-melanoma skin cancers or cancers that have clearly been cured or in the option of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer)
* Have autoimmune or collagen vascular diseases
* Have immunodeficiency diseases or HIV
* You have any other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator are life-threatening or that may interfere with study participation or the ability to follow the intervention protocol.

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-12; Primary Completion 2015-07 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Newton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Newton RL Jr, Johnson WD, Hendrick C, Harris M, Andrews E 3rd, Johannsen N, Rodarte RQ, Hsia DS, Church TS. A randomized controlled exercise training trial on insulin sensitivity in African American men: The ARTIIS study: Major category: study design, statistical design, study protocols. Contemp Clin Trials. 2015 Jul;43:75-82. doi: 10.1016/j.cct.2015.05.004. Epub 2015 May 12. PMID 25979318
- [Background] Newton RL Jr, Johnson WD, Larrivee S, Hendrick C, Harris M, Johannsen NM, Swift DL, Hsia DS, Church TS. A Randomized Community-based Exercise Training Trial in African American Men: Aerobic Plus Resistance Training and Insulin Sensitivity in African American Men. Med Sci Sports Exerc. 2020 Feb;52(2):408-416. doi: 10.1249/MSS.0000000000002149. PMID 31939911

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Started | 56 | 57
Completed | 54 | 51
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Aerobic Plus Resistance Training Group | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 55 | 106
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (8.13) | 50.54 (9.59) | 51.99 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 56 | 57 | 113
Region of Enrollment [Number; unit: participants]
  United States | 56 | 57 | 113

OUTCOME MEASURES:

1. Primary Outcome: Insulin Response to an Oral Glucose Tolerance Test Over 20 Weeks.
Description: An oral glucose tolerance test is a medical test in which glucose is given and blood samples are taken afterward to determine how quickly it is cleared from the blood. The test is usually used to test for diabetes or insulin resistance.
Time Frame: Baseline, week 10, week 20
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: uU/mL
Groups:
- Control Group: We will randomly assign 56 individuals to a no exercise healthy living group.
  Control Group: Participants randomized into the control group will not be provided with memberships to any exercise facility, nor will they receive behavioral instruction on how to increase physical activity. They will receive information on living a healthy lifestyle. Such minimal interventions have not been shown to increase physical activity in participants. The participants in this group will undergo the baseline, 10 week, and 20 week testing.
- Aerobic Plus Resistance Training Group: We will randomly assign 57 individuals to an aerobic plus resistance training group.
  Aerobic Plus Resistance Training Group: Participants randomized to this intervention will engage in both aerobic and resistance training in accordance with Physical Activity Guidelines for Americans, that is 150 minutes of aerobic training and 2 days of additional 20 minutes of resistance training. The aerobic training component will be completed on a treadmill and target training intensity will be self-selected at 65% to 85% of maximal aerobic capacity. Each resistance training session will consist of both upper and lower body exercises: 2 sets of 9 exercises with each set consisting of 10 repetitions.
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
uU/mL
  Baseline | 110.51 (8.14) | 106.64 (7.77)
  Week 10: number analyzed (Participants) | 49 | 54
  Week 10 | 90.68 (8.13) | 80.23 (6.52)
  Week 20: number analyzed (Participants) | 49 | 54
  Week 20 | 86.7 (7.3) | 80.74 (7.25)

2. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure was measured at rest using a standard mercury sphygmomanometer.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
mmHg
  Baseline | 81.2 (1.04) | 81.74 (1.16)
  Week 10: number analyzed (Participants) | 47 | 52
  Week 10 | 72.13 (1.04) | 70.8 (1.06)
  Week 20: number analyzed (Participants) | 47 | 52
  Week 20 | 79.16 (1.09) | 79.85 (1.27)

3. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured at rest using a standard mercury sphygmomanometer.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Control Group: We will randomly assign 56 individuals to a no exercise healthy living group.
  Control Group: Participants randomized into the control group will not be provided with memberships to any exercise facility, nor will they receive behavioral instruction on how to increase physical activity. They will receive information on living a healthy lifestyle. Such minimal interventions have not been shown to increase physical activity in participants.
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
mm Hg
  Baseline | 123.04 (1.5) | 124.39 (1.62)
  Week 10: number analyzed (Participants) | 47 | 52
  Week 10 | 116.13 (1.53) | 114.84 (1.64)
  Week 20: number analyzed (Participants) | 47 | 52
  Week 20 | 120.06 (1.6) | 122.68 (1.76)

4. Secondary Outcome: Body Composition
Description: Body composition was assessed using the General Electric (General Electric; Milwaukee, WI) Lunar i-Dual energy X-ray absorptiometry.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
kg
  Baseline | 100.79 (2.54) | 99.75 (2.25)
  Week 20: number analyzed (Participants) | 49 | 54
  Week 20 | 99.46 (2.82) | 97.97 (2.39)

5. Secondary Outcome: Cardiorespiratory Fitness
Description: Fitness testing is being used as a measure of change in the aerobic component of the intervention. Cardiorespiratory fitness maximal exercise tests were conducted using a standardized graded exercise testing protocol administered on a treadmill.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: L/min of oxygen
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
L/min of oxygen
  Baseline | 2.41 (0.07) | 2.41 (0.07)
  Week 20: number analyzed (Participants) | 44 | 44
  Week 20 | 2.3 (0.09) | 2.6 (0.09)

6. Secondary Outcome: Muscular Strength
Description: Strength testing is performed in order to assess change in response to the resistance training program. Muscular strength is measured via isokinetic testing on a Biodex System 4 Isokinetic Dynamometer.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: Joules
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
Joules
  Baseline | 3926.1 (788.2) | 4011.0 (833.2)
  Week 20: number analyzed (Participants) | 45 | 43
  Week 20 | 3999.5 (984.3) | 4113.7 (972.3)

7. Secondary Outcome: Mood
Description: Depressive symptomatology is measured by the Center for Epidemiology Studies Depression Scale (CES-D). The total score range is 0 to 60. Higher scores represent higher levels of depressive symptomatology.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
score on a scale
  Baseline | 5.75 (0.59) | 6.05 (0.66)
  Week 20: number analyzed (Participants) | 49 | 54
  Week 20 | 10.09 (0.99) | 10.37 (1.04)

8. Secondary Outcome: Mental Health
Description: The Health Related Quality of Life (SF-36) questionnaire is being used to assess perceived quality of life, which usually improves through regular exercise. The measure is scored on a T-scale, with a mean of 50 and standard deviation of 10. Higher scores represent better functioning. Scores below 40 suggest poorer functioning than normal, and scores above 60 represent better functioning than normal.
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
T-score
  Baseline | 56.59 (0.85) | 55.53 (0.89)
  Week 20: number analyzed (Participants) | 55 | 57
  Week 20 | 57.27 (0.71) | 54.41 (1.21)

9. Secondary Outcome: Physical Health
Description: as for outcome 8
Time Frame: 20 weeks
Population: The number analyzed differs by row because some participants did not complete the follow-up measures.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Control Group | Aerobic Plus Resistance Training Group
Number analyzed (Participants) | 56 | 57
T-score
  Baseline | 55.84 (0.51) | 55.35 (0.8)
  Week 20: number analyzed (Participants) | 55 | 57
  Week 20 | 54.96 (0.79) | 53.4 (1.11)

ADVERSE EVENTS:
Groups:
- Healthy Living Control: Participants assigned to the Healthy Living Group will receive health information through newsletters via email or standard mail throughout the study. They will also receive a monthly phone call from the coordinator to assess their current health status and capture any adverse events that have occurred within that month. We have found that participants assigned to these health information control groups report being satisfied with the information and their assignment. Monthly newsletters issued to participants in this group will feature such things as nutrition articles, healthy recipes, and diabetes education. We will focus heavily on diabetes education and prevention. Participants will be asked to complete satisfaction surveys throughout the intervention. After the five month intervention is complete, participants will be given a 5 month membership to the YMCA. Attendance to the YMCA will be verified via card scan reports throughout the duration of the study.
- Aerobic Plus Resistance Training Group: Participants randomized to this intervention will engage in both aerobic and resistance training in accordance with Physical Activity Guidelines for Americans, that is 150 minutes of aerobic training and 2 days of an additional 20-30 minutes of resistance training. The intervention lasts 5 months. The resistance training regimen will remain constant at 2 days per week, for 20-30 minutes, regardless of the number of days of aerobic training. Each resistance training session will consist of 2 sets of 9 exercises with each set consisting of 10-12 repetitions. Therefore, the circuit resistance machines to be used in the study are the abdominal crunch, vertical chest press, shoulder press, leg press, leg extension, and leg curl. Resistance will be increased when an individual can comfortably perform 10 repetitions of the exercise.
Arm/Group | Healthy Living Control | Aerobic Plus Resistance Training Group
Serious Adverse Events (participants affected / at risk) | 0/56 | 1/57
Other Adverse Events (participants affected / at risk) | 4/56 | 16/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Living Control (N=56) | Aerobic Plus Resistance Training Group (N=57)
Illness (Skin and subcutaneous tissue disorders) | 0 | 1 — Hospitalized overnight for a boil.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Living Control (N=56) | Aerobic Plus Resistance Training Group (N=57)
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 1 | 0 — Bursitis in hip.
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 1 | 0 — L Achilles tear, surgical repair secondary to a fall at work.
Abnormal lab values (General disorders) | 1 | 0 — Diagnosed with T2DM.
Muscle/Joint/Injury (Hepatobiliary disorders) | 1 | 0 — Sprained L knee refereeing basketball game
Muscle/Joint/Injury (Renal and urinary disorders) | 0 | 1 — Prostate resection surgery.
Muscle/Joint/Injury (Renal and urinary disorders) | 0 | 1 — Prostate procedure (h/o BPH).
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Muscle spasms secondary to MVA
Surgery/hospitalization (Musculoskeletal and connective tissue disorders) | 0 | 1 — Left shoulder pain.
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Neck pain secondary to MVA.
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Shoulder strain secondary to fall on treadmill during intervention.
Abnormal lab values (Musculoskeletal and connective tissue disorders) | 0 | 1 — Back pain.
Surgery/hospitalization (Musculoskeletal and connective tissue disorders) | 0 | 1 — L knee strain at work.
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — L shoulder pain (prior history)
Muscle/Joint/Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — L shoulder pain after sleeping funny.
GI (Musculoskeletal and connective tissue disorders) | 0 | 1 — Lower back pain & R lower extremity pain secondary to MVA.
Illness (Gastrointestinal disorders) | 0 | 1 — Stomach pain, missed intervention for 1 week.
Hypoglycemia (Endocrine disorders) | 0 | 1 — Abnormal thyroid test.
Surgery/hospitalization (Nervous system disorders) | 0 | 1 — Recurrent headaches.
Muscle/Joint/Injury (General disorders) | 0 | 1 — Flu.
Muscle/Joint/Injury (General disorders) | 0 | 1 — Nausea & weakness during exercise (no breakfast)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes